CLINICAL TRIAL: NCT01226680
Title: A Phase II, Randomized, Double Masked, Parallel Group, Vehicle Controlled, Multiple-Dose Study Of Tasocitinib (CP-690,550) In Subjects With Dry Eye Disease
Brief Title: A Study Of Tasocitinib In Dry Eye Subjects
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3921066
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Keratoconjunctivitis Sicca
Keywords: Dry Eye; Schirmer test; corneal staining; OSDI; OCI
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tasocitinib 0.005% QD (Experimental)
  Interventions: Drug: Tasocitinib
- Tasocitinib 0.003% QD (Experimental)
  Interventions: Drug: Tasocitinib
- Vehicle for Tasocitinib (Placebo Comparator)
  Interventions: Drug: vehicle for Tasocitinib

INTERVENTIONS:
Drug: Tasocitinib — 0.005% QD for 12 weeks
  Arms: Tasocitinib 0.005% QD
Drug: Tasocitinib — 0.003% QD for 12 weeks
  Arms: Tasocitinib 0.003% QD
Drug: vehicle for Tasocitinib — vehicle QD for 12 weeks
  Arms: Vehicle for Tasocitinib

SUMMARY:
This is a phase 2 study to further evaluate the safety and efficacy of tasocitinib (CP-690,550) in the subjects with moderate to severe dry eye disease. Both subjective and objective clinical endpoints will be measured for a duration of 12-week treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 years or older at time of consent
* Diagnosis of dry eye disease, characterized by subjective symptoms of dry eye for at least 6 months, Schirmer test without anesthesia: =>1 mm and =<7 mm, sum of corneal fluorescein staining score of =>4 (NEI Scale), and subject grading total score of => 23 on the OSDI

Exclusion Criteria:

* Planned initiation of, or changes to, concomitant medication that could affect dry eye within 30 days of the Screening visit or during study
* Ocular disorders that may confound interpretation of study results such as significant corneal surface disease not caused by dry eyes, abnormal corneal sensitivity, abnormal tear spreading, including but not limited to the following: abnormal lid function, lid position, or blink rate, that in the opinion of the investigator is clinically significant, history of herpetic keratopathy
* Lacrimal punctal occlusion (plugs or cautery) within 2 months of the Screening visit
* Contact lens wear within 2 weeks of the Screening visit and/or during study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12-01 (Actual); Primary Completion 2012-10-19 (Estimated); Study Completion 2012-10-19 (Estimated)

PRIMARY OUTCOMES:
Change in length of wetting of Schirmer test strip without anesthesia from baseline | Week 12
Change in Ocular Surface Disease Index's Environmental Trigger (OSDI-ET) subscale score from baseline | Week 12

SECONDARY OUTCOMES:
Systemic safety: adverse events, clinical laboratory; and vital signs | 12 weeks
Ocular tolerability and safety: incidence and severity of ocular adverse events during the study (ophthalmic examination, ocular tolerability assessment and/ or adverse events spontaneously reported) | 12 weeks
Schirmer test without anesthesia: Change in length of wetting from baseline at Days 7, 14, 28, and Week 8; Response rate (percentage of subjects who achieve ≥10mm wetting) at Days 7, 14, 28, and Weeks 8 and 12; Response rate (percentage of | 12 weeks
subjects who achieve increase of ≥10mm wetting) at Days 7, 14, 28, and Weeks 8 and 12; Time to achievement of change from baseline of ≥10mm wetting;Time to achievement of ≥10mm wetting | 12 weeks
Corneal staining:Change from baseline at Days 7, 14, 28 and Weeks 8 and 12;Response rate (percentage of subjects who demonstrate 100% clearing of corneal staining) at Days 7, 14, 28 and Weeks 8 and 12;Time to achievement of 100% clearing of corneal | 12 weeks
staining | 12 weeks
Ocular Surface Disease Index (OSDI): Change in the OSDI total score and three subscale scores (the Ocular Symptoms, Vision-Related Function, and Environmental Triggers) from baseline at Days 7, 14, 28, and Weeks 8 and 12 (except ET subscale | 12 weeks
score); Response rate (percentage of subjects who demonstrating ≥10 unit decrease in OSDI total score) at Days 7, 14, 28, and Weeks 8 and 12; Time to achievement of ≥10 unit decrease in OSDI total score | 12 weeks
Modified Ocular Comfort Index (mOCI): Change in the OCI score, the Dry Eye Symptoms (DES) and Symptom Interference (SI) subscales scores from baseline at Days 7, 14, 28 and Weeks 8 and 12; OCI Response rate (percentage of subjects who demonstrating | 12 weeks
≥3 point decrease from baseline in the OCI score) at Days 7, 14, 28, and Weeks 8 and 12; Time to achievement of ≥3 point decrease from baseline in the OCI score | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921066&StudyName=A%20Study%20Of%20Tasocitinib%20In%20Dry%20Eye%20Subjects